CLINICAL TRIAL: NCT00072046
Title: A Randomized Phase III Trial Of Interferon Alfa-2B Or Interferon Alfa-2B Plus Bevacizumab In Patients With Advanced Renal Carcinoma
Brief Title: Interferon Alfa-2b With or Without Bevacizumab in Treating Patients With Advanced Renal Cell Carcinoma (Kidney Cancer)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-90206; U10CA031946 (NIH); CAN-NCIC-REC1; CDR0000335292 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; clear cell renal cell carcinoma; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Bevacizumab; Interferon-alpha

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interferon (Experimental): Treatment with interferon alfa 2b
  Interventions: Biological: recombinant interferon alfa
- Interferon + bevacizumab (Experimental): Addition of bevacizumab to interferon alfa 2b treatment
  Interventions: Biological: bevacizumab; Biological: recombinant interferon alfa

INTERVENTIONS:
Biological: bevacizumab — 10mg/kg IV infusion on Days 1 & 15 of each cycle
  Arms: Interferon + bevacizumab
Biological: recombinant interferon alfa — 9 million units subQ injection 3 x/week for 4 weeks

SUMMARY:
RATIONALE: Biological therapies, such as interferon alfa-2b, may interfere with the growth of tumor cells. Bevacizumab may stop the growth of tumor cells by stopping blood flow to the tumor. It is not yet known whether interferon alfa-2b is more effective with or without bevacizumab in treating advanced renal cell carcinoma (kidney cancer).

PURPOSE: This randomized phase III trial is studying interferon alfa-2b and bevacizumab to see how well they work compared to interferon alfa-2b alone in treating patients with advanced renal cell carcinoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival of patients with advanced renal cell carcinoma treated with interferon alfa-2b alone or interferon alfa-2b with bevacizumab.

Secondary

* Compare the time to disease progression and objective response rates in patients treated with these regimens.
* Determine the toxicity of interferon alfa-2b in combination with bevacizumab in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prior nephrectomy (yes vs no) and number of risk factors for disease progression (0 vs 1-2 vs 3 or more). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive interferon alfa-2b subcutaneously (SC) three times a week.
* Arm II: Patients receive interferon alfa-2b as in arm I and bevacizumab IV over 30-90 minutes on days 1 and 15.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then annually for up to 10 years after study entry.

PROJECTED ACCRUAL: A total of 700 patients (350 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed renal cell carcinoma (RCC)

  * Conventional clear cell carcinoma
  * Metastatic or unresectable disease
* The following characteristics and cellular types are excluded:

  * True papillary
  * Sarcomatoid features without a clear cell component
  * Chromophobe
  * Oncocytoma
  * Collecting duct tumor
  * Transitional cell carcinoma
* Measurable or nonmeasurable disease, including any of the following:

  * Unidimensionally measurable lesion ≥ 20 mm by conventional techniques (e.g., physical exam or chest x-ray) OR 10 mm by spiral CT scan or MRI
  * The following are considered nonmeasurable disease:

    * Small lesions
    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
    * Irradiated lesions, unless progression is documented after radiotherapy
* RCC paraffin tissue blocks or unstained slides must be available
* No evidence of prior or concurrent CNS metastases by MRI or CT scan

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No history of clinically significant bleeding

Hepatic

* AST/ALT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin ≤ 1.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN
* No proteinuria > 1+

  * Proteinuria ≥ 2+ allowed provided protein is < 2 g/24-hour urine collection

Cardiovascular

* No deep venous thrombosis within the past year
* No cerebrovascular accident within the past year
* No peripheral vascular disease with claudication on < 1 block
* No uncontrolled hypertension defined as blood pressure ≥160 mm Hg (systolic) and/or ≥ 90 mm Hg (diastolic) while on medication
* No New York Heart Association class II-IV congestive heart failure
* No angina pectoris requiring nitrate therapy
* No myocardial infarction within the past 6 months
* No other significant cardiovascular disease

Pulmonary

* No pulmonary embolus within the past year
* No ongoing hemoptysis

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study treatment
* No preexisting thyroid abnormality in which normal thyroid function cannot be maintained by medication
* No delayed wound healing, ulcers, or bone fractures
* No uncontrolled psychiatric disorder
* No other currently active* malignancy except nonmelanoma skin cancer NOTE: *Disease is not considered currently active if patient completed anticancer therapy and is considered to have < 30% risk of relapse

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior systemic immunotherapy for RCC
* No prior thalidomide, anti-vascular endothelial growth factor (VEGF) therapy, VEGF receptor inhibitors, or antiangiogenic treatment of any kind
* No concurrent prophylactic filgrastim (G-CSF) or sargramostim (GM-CSF)

Chemotherapy

* No prior systemic chemotherapy for RCC
* No concurrent chemotherapy

Endocrine therapy

* No concurrent systemic corticosteroid therapy except the following:

  * Topical and inhaled steroids
  * Replacement therapy for adrenal insufficiency
* No concurrent hormones except those administered for nondisease-related conditions (e.g., insulin for diabetes)

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* Prior palliative radiotherapy to metastatic lesions allowed provided at least 1 measurable or nonmeasurable lesion remains untreated
* No concurrent palliative radiotherapy

Surgery

* At least 4 weeks since prior major surgery and recovered

Other

* No other prior systemic investigational therapy for RCC
* No other prior adjuvant or neoadjuvant systemic therapy for RCC
* No concurrent full-dose oral or parenteral anticoagulation* NOTE: *Low-dose (1 mg) warfarin for maintenance of catheter patency and/or daily prophylactic aspirin is allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 732 (Actual)
Dates: Start 2003-10; Primary Completion 2004-01 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 5 years

SECONDARY OUTCOMES:
Time to progression | q 3 cycles
Toxicity | q cycle

CONTACTS AND LOCATIONS:
Overall Officials: Brian I. Rini, MD, Study Chair — University of California, San Francisco
Locations (493):
- United States (489):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Huntsville Hospital, Huntsville, Alabama
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Arroyo Grande Community Hospital, Arroyo Grande, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Providence Holy Cross Cancer Center, Mission Hills, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Rebecca and John Moores UCSD Cancer Center, San Diego, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Naval Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - San Francisco General Hospital Medical Center, San Francisco, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Cancer Center of Colorado Springs, Colorado Springs, Colorado
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thorton, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Middlesex Hospital Cancer Center, Middletown, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Kent General Hospital at Bayhealth Medical Center, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - St. Francis Hospital, Wilmington, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Lynn Regional Cancer Center of Boca Raton Community Hospital, Boca Raton, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Shands Cancer Center at the University of Florida - Jacksonville, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - Watson Clinic, Lakeland, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Oncology Associates, Orange Park, Florida
  - Florida Hospital - Orlando, Orlando, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Palm Beach Cancer Institute - West Palm Beach, West Palm Beach, Florida
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - Emory University Hospital - Atlanta, Altanta, Georgia
  - Hematology and Oncology of Northeast Georgia, Athens, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Augusta Oncology Associates, Augusta, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B. Amos Community Cancer Center, Columbus, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Care and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolula, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - St. Francis Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Mountain States Tumor Institute - Boise, Boise, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Illinois Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Alexian Brothers Cancer Care Center, Elk Grove Village, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Evanston Northwestern Health Care - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Medical and Surgical Specialists, LLC, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology Hematology Associates, Limited - West, Joliet, Illinois
  - Provena St. Mary's Wasser Regional Cancer Center - Kankakee, Kankakee, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Medical Center - East, Moline, Illinois
  - Hematology Oncology Consultants Ltd., Naperville, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Oncology Institute of Greater Lafayette, Lafayette, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Saint Joseph Regional Medical Center - Plymouth Campus, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McFarland Clinic, P.C., Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Wendt Regional Cancer Center at Finley Hospital, Dubuque, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Alegent Health Community Memorial Hospital, Missouri Valley, Iowa
  - Burgess Health Center, Onawa, Iowa
  - Cancer Center at Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Mount Carmel Regional Cancer Center, Pittsburg, Kansas
  - Pratt Cancer Center of Kansas, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center at Stormont-Vail Regional Health Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates in Womens Health, Wichita, Kansas
  - Cancer Center of Kansas, P.A., Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baton Rouge General Regional Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Clinic of Baton Rouge, Baton Rouge, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Cancer Center at Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - St. Agnes Cancer Center, Baltimore, Maryland
  - Union Hospital Cancer Center at Union Hospital, Elkton MD, Maryland
  - Cancer Center at Tufts - New England Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Commonwealth Hematology-Oncology P.C. - Quincy, Quincy, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Battle Creek Health System, Battle Creek, Michigan
  - Mecosta County General Hospital, Big Rapids, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Mercy Medical Center, Grand Rapids, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Metropolitan Hospital, Grand Rapids, Michigan
  - Spectrum Health Hospital - Blodgett Campus, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Foote Hospital, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, P.C., Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - Oncology Care Associates, P.L.L.C., Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Brainerd Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Cancer Care Center at St. Luke's Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Mercy and Unity Hospitals, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Adult and Pediatric Urology, P.L.L.P., Saint Cloud, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Clinic, Saint Louis Park, Minnesota
  - Cancer Care Center at Regions Hospital, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Woodwinds Hospital, Woodbury, Minnesota
  - Hematology & Oncology Clinic, Hattiesburg, Mississippi
  - Hattiesburg Clinic, P.A., Hattiesburg, Mississippi
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - St. Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Missouri Cancer Associates, Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Freeman Cancer Institute at Freeman Health System, Joplin, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - St. Anthony's Cancer Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - Fremont Area Medical Center, Fremont, Nebraska
  - Cancer Center at the Good Samaritan Health Systems, Kearney, Nebraska
  - Bryan LGH Medical Center West, Lincoln, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - St. Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - Alegent Health - Immanuel Medical Center, Omaha, Nebraska
  - Bergan Mercy Medical Center, Omaha, Nebraska
  - Cancer Center at Creighton University Medical Center, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Cancer Center at Midlands Community Hospital, Papillion, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Washoe Cancer Services at Washoe Medical Center - Reno, Reno, Nevada
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Frisbie Memorial Hospital, Rochester, New Hampshire
  - Cancer Institute of New Jersey at the Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Cancer Center at the Mountainside Hospital, Montclair, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Warren Hospital, Phillipsburg, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Hematology-Oncology Associates, PC, Albuquerque, New Mexico
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Lovelace Medical Center at Lovelace Sandia Health System, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Louis Busch Hager Cancer Center at Mary Imogene Bassett Hospital, Cooperstown, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Beth Israel Medical Center - Petrie Division, New York, New York
  - St. Luke's-Roosevelt Hospital Center - St.Luke's Division, New York, New York
  - Union State Bank Cancer Center at Nyack Hospital, Nyack, New York
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - St. Joseph's Hospital Health Center - Syracuse, Syracuse, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Comprehensive Cancer Center at Our Lady of Mercy Medical Center, The Bronx, New York
  - Faxton Regional Cancer Center, Utica, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - John Smith, Jr./Dalton McMichael Cancer Center at Morehead Memorial Hospital, Eden, North Carolina
  - Comprehensive Cancer Center at Gaston Memorial, Gastonia, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Leo W. Jenkins Cancer Center at Pitt County Memorial Hospital, Greenville, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Health System, Bismarck, North Dakota
  - Mid Dakota Clinic, P.C., Bismarck, North Dakota
  - Dakota Cancer Institute at Innovis Health - Dakota Clinic, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron City Hospital at Summa Health System, Akron, Ohio
  - St. Elizabeth Boardman Cancer Center, Boardman, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - University Hospitals Ireland Cancer Center at Mercy Medical Center, Canton, Ohio
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Kenton Oncology, Inc., Kenton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center Oncology Unit, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Promedica Cancer Center at Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical College of Ohio Cancer Institute, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated, Toledo, Ohio
  - Toledo Surgical Specialists, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - St. Joseph Health Care Center, Warren, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - United States Air Force Medical Center Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - St. Elizabeth Cancer Center at St. Elizabeth Health Center - Youngstown, Youngstown, Ohio
  - Comanche County Memorial Hospital, Lawton, Oklahoma
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Mercy Health Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - John and Dorothy Morgan Cancer Center at Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, P.C. at Hahne Regional Cancer Center, DuBois, Pennsylvania
  - PinnacleHealth Regional Cancer Center at Polyclinic Hospital, Harrisburg, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Central Pennsylvania Hematology and Medical Oncology Associates, PC, Lemoyne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Guthrie Medical Center - Sayre, Sayre, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital at Lifespan, Providence, Rhode Island
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Jones Clinic, Germantown, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Baptist Hospital Of East Tennessee, Knoxville, Tennessee
  - Arlington Cancer Center - Arlington, Arlington, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Virginia Oncology Associates - Hampton, Hampton, Virginia
  - Rappahannock General Hospital, Kilmarnock, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Providence Cancer Center at Holy Family Hospital, Spokane, Washington
  - North Star Lodge Cancer Center, Yakima, Washington
  - Washington Hematology - Oncology Specialists, Yakima, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Marshall University Medical Center, Huntington, West Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Fox Valley Hematology and Oncology, Appleton, Wisconsin
  - Vince Lombardi Cancer Center - Elkhorn, Elkhorn, Wisconsin
  - Oncology Alliance, S.C. - Milwaukee - East, Glendale, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - UW Health Oncology, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center, Manitowoc, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Medical Consultants, Milwaukee, Wisconsin
  - Froedtert Hospital and Medical College of Wisconcin, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - All Saints Cancer Center at All Saints Healthcare, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic - Sheboygan, Sheboygan, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - University of Wisconsin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
- Canada (4):
  - University of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Nova Scotia Cancer Centre at Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan

REFERENCES:
- [Result] Rini BI, Halabi S, Rosenberg JE, Stadler WM, Vaena DA, Archer L, Atkins JN, Picus J, Czaykowski P, Dutcher J, Small EJ. Phase III trial of bevacizumab plus interferon alfa versus interferon alfa monotherapy in patients with metastatic renal cell carcinoma: final results of CALGB 90206. J Clin Oncol. 2010 May 1;28(13):2137-43. doi: 10.1200/JCO.2009.26.5561. Epub 2010 Apr 5. PMID 20368558
- [Result] Rini BI, Halabi S, Rosenberg J, et al.: Bevacizumab plus interferon-alpha versus interferon-alpha monotherapy in patients with metastatic renal cell carcinoma: results of overall survival for CALGB 90206. [Abstract] J Clin Oncol 27 (Suppl 15): A-LBA5019, 2009.
- [Result] Rini BI, Halabi S, Rosenberg JE, et al.: CALGB 90206: a phase III trial of bevacizumab plus interferon-alpha versus interferon-alpha monotherapy in metastatic renal cell carcinoma. [Abstract] American Society of Clinical Oncology 2008 Genitourinary Cancers Symposium, Feb 14-16, 2008, San Francisco, CA. A-350, 2008.
- [Result] Rini BI, Halabi S, Rosenberg JE, Stadler WM, Vaena DA, Ou SS, Archer L, Atkins JN, Picus J, Czaykowski P, Dutcher J, Small EJ. Bevacizumab plus interferon alfa compared with interferon alfa monotherapy in patients with metastatic renal cell carcinoma: CALGB 90206. J Clin Oncol. 2008 Nov 20;26(33):5422-8. doi: 10.1200/JCO.2008.16.9847. Epub 2008 Oct 20. PMID 18936475
- [Result] Rini BI, Halabi S, Taylor J, Small EJ, Schilsky RL; Cancer and Leukemia Group B. Cancer and Leukemia Group B 90206: A randomized phase III trial of interferon-alpha or interferon-alpha plus anti-vascular endothelial growth factor antibody (bevacizumab) in metastatic renal cell carcinoma. Clin Cancer Res. 2004 Apr 15;10(8):2584-6. doi: 10.1158/1078-0432.ccr-03-0605. PMID 15102658
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Nixon AB, Halabi S, Liu Y, Starr MD, Brady JC, Shterev I, Luo B, Hurwitz HI, Febbo PG, Rini BI, Beltran H, Small EJ, Morris MJ, George DJ. Predictive Biomarkers of Overall Survival in Patients with Metastatic Renal Cell Carcinoma Treated with IFNalpha +/- Bevacizumab: Results from CALGB 90206 (Alliance). Clin Cancer Res. 2022 Jul 1;28(13):2771-2778. doi: 10.1158/1078-0432.CCR-21-2386. PMID 34965953